CLINICAL TRIAL: NCT05672706
Title: A Study of Pressure Waveform Analysis in Coronary Artery-II
Status: Recruiting | Type: Observational
Sponsor: National Taiwan University Hospital Hsin-Chu Branch (Other)
Responsible Party: Sponsor
Other Study IDs: 111-129-E
Record Dates: First submitted 2023-01-03; First posted 2023-01-05 (Actual); Last update posted 2023-01-05 (Actual); Status verified 2023-01

CONDITIONS: Ischemic Heart Disease
MeSH Terms: conditions — Myocardial Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples Without DNA — 4ml serum was collected at the end of the FFR procedure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CFR and IMR group
  Interventions: Procedure: CFR and IMR group

INTERVENTIONS:
Procedure: CFR and IMR group — Participants will undergo repeat intracoronary adenosine administration during CFR and IMR measurement

SUMMARY:
The goal of this observational study is to test the feasibility of intracoronary adenosine administration during coronary flow reserve(CFR) and index of microcirculatory resistance(IMR) assessment in a population with angina. The main questions it aims to answer are:

* Repeatability of CFR and IMR assessment while hyperemia with intracoronary adenosine was administered.
* Evaluate the correlation of the intrinsic signal of coronary waveform versus physiologic ischemia, while defined by fractional flow reserve(FFR) and CFR respectively.
* The predictive value of FFR, CFR, and IMR on major adverse cardiovascular outcomes in 3 years Participants will undergo FFR, CFR, and IMR assessments in the catheterization laboratory of the National Taiwan University Hospital Hsin-Chu Branch, then clinical events follow up for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Participants with angina

Exclusion Criteria:

* Severe valvular heart disease
* History of asthma
* Heart rate less than 50 beats per minute
* systolic blood pressure less than 90 mmHg

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with angina and undergo invasive coronary angiography
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-01-04 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Repeatability of CFR and IMR value | 10 minutes
  To compare the difference of individual value, while repeat the measurement within 1 minutes

SECONDARY OUTCOMES:
Major adverse cardiovascular outcomes | 3 year
  Including death, myocardial infarction, stroke and heart failure

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital Hsin-Chu branch, Hsinchu, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided